CLINICAL TRIAL: NCT00712920
Title: Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of MP03-36 and MP03-33 in Patients With Perennial Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Nasal Spray to Treat Perennial Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Harry Sacks, MD Vice President, Medical and Scientific Affairs, Meda Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP434
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Results first posted 2010-01-15 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): 0.15% azelastine hydrochloride 1644 mcg/2 sprays per nostril 2 times a day for 4 weeks
  Interventions: Drug: 0.15% azelastine hydrochloride
- 3 (Experimental): 0.1% azelastine hydrochloride 1096 mcg/2 sprays per nostril 2 times a day for 4 weeks
  Interventions: Drug: 0.1% azelastine hydrochloride

INTERVENTIONS:
Drug: 0.15% azelastine hydrochloride — 0.15% azelastine hydrochloride 1644 mcg
  Arms: 2
Drug: 0.1% azelastine hydrochloride — 0.1% azelastine hydrochloride 1096 mcg
  Arms: 3
Drug: Placebo — Placebo
  Arms: 1

SUMMARY:
The purpose of this study is to determine if two allergy medications are more effective than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 12 years of age and older
* Must be in generally good health
* Must meet minimum symptom requirements, as specified in protocol
* Must be willing and able to provide informed consent and participate in all study procedures
* 2-year history of PAR
* Positive skin test to cockroach, dust mite, mold or cat/dog dander

Exclusion Criteria:

* On nasal examination, presence of any nasal mucosal erosion, nasal ulceration or nasal septal perforation at the screening or randomization visit
* Nasal diseases likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa, significant polyposis or nasal structural abnormalities
* Nasal surgery or sinus surgery within the previous year
* The use of any investigational drug within 30 days
* Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose
* Women who are pregnant or nursing
* Women of child-bearing potential who are not abstinent and not practicing a medically acceptable method of contraception
* Respiratory tract infection within 2 weeks of screening
* Respiratory tract infections requiring oral antibiotic treatment within 2 weeks of screening
* Patients with asthma with the exception of mild, intermittent
* Significant pulmonary disease including COPD
* Patients with arrhythmia
* Patients with a known history of alcohol or drug abuse
* Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor may significantly alter the absorption, distribution, metabolism or excretion of study drug.
* Clinically relevant abnormal physical findings within one week of randomization
* Overnight abscences from home for more than 3 nights
* Employees of the research center or private practice and family members are excluded
* Patients who received prohibited medications within specified timepoints in protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Allergy and Asthma Specialist Medical Group, Huntington Beach, California
  - Allergy, Asthma and Respiratory Care medical Center, Long Beach, California
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Allergy Associates Medical Group Inc, San Diego, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - Asthma and Allergy Associates, Colorado Springs, Colorado
  - The William Storms Allergy Clinic, Colorodo Springs, Colorado
  - Atlanta Allergy and Asthma Clinic, Woodstock, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - Institute for Asthma and Allergy PC, Wheaton, Maryland
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Las Vegas Physicians Research Group, Henderson, Nevada
  - Allergy and Asthma Research NJ inc, Mount Laurel, New Jersey
  - Atlantic Research Center, Ocean City, New Jersey
  - Dr. Perin, Teaneck, New Jersey
  - AAIR Research Center, Rochester, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - New Horizon's Clinical Research, Cincinnati, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy Asthma and Dermatology Research, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy and Consultants of NJ/PA, Collegeville, Pennsylvania
  - Asthma and Allergy Research Associate, Upland, Pennsylvania
  - Asthma, Nasal Disease & Allergy Research Center of New England, Providence, Rhode Island
  - National Allergy, Asthma and Urticaria of Charleston, Charleston, South Carolina
  - Allergy and Asthma Associates, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Pharmaceutical Research & Consulting Inc, Dallas, Texas
  - Central Texas Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy and Asthma Center, Waco, Texas
  - Virginia Adult & Pediactric Allergy & Asthma, PC, Richmond, Virginia
  - Asthma, Inc., Seattle, Washington
  - Advanced Healthcare, SC, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Bousquet J, Klimek L, Kuhl HC, Nguyen DT, Ramalingam RK, Canonica GW, Berger WE. A double-blind, placebo-controlled trial of the efficacy and safety of two doses of azelastine hydrochloride in perennial allergic rhinitis. Front Allergy. 2023 Oct 18;4:1244012. doi: 10.3389/falgy.2023.1244012. eCollection 2023. PMID 37920410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Observation: February 5, 2007 Last Observation: October 8, 2007
Pre-assignment Details: Subjects participated in a 7 day screening period to Identify appropriate subjects based on symptom scores.
Groups:
- Placebo: Placebo nasal Spray/2 sprays per nostril 2 times a day for 4 weeks
- Astepro 0.1%: 0.10% azelastine hydrochloride 1096 mcg nasal Spray/2 sprays per nostril 2 times a day for 4 weeks
- Astepro 0.15%: 0.15% azelastine hydrochloride 1644 mcg nasal Spray/2 sprays per nostril 2 times a day for 4 weeks
Period: Overall Study
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Started | 192 | 197 (3 subjects were randomized in error) | 192
Completed | 175 | 180 | 180
Not Completed | 17 | 17 | 12
Not completed — Adverse Event | 3 | 4 | 7
Not completed — Withdrawal by Subject | 4 | 2 | 1
Not completed — Lost to Follow-up | 1 | 4 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Other | 5 | 7 | 3
Not completed — Non-compliance | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15% | Total
Number analyzed (Participants) | 192 | 194 | 192 | 578
Age, Categorical [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    <=18 years | 21 | 11 | 18 | 50
    Between 18 and 65 years | 161 | 183 | 170 | 514
    >=65 years | 10 | 0 | 4 | 14
Age Continuous [Mean (Standard Deviation); unit: years] — Number of participants based on ITT population
  years | 38.1 (15.37) | 36.9 (13.09) | 35.6 (13.31) | 36.9 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    Female | 130 | 136 | 127 | 393
    Male | 62 | 58 | 65 | 185
Region of Enrollment [Number; unit: participants] — Number of participants based on ITT population
  participants
    United States | 192 | 194 | 192 | 578

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-hour Reflective Total Nasal Symptom Score (AM and PM Combined) at 28 Days.
Description: Reflective total nasal symptom score consisting of Runny nose, itchy nose, nasal Congestion, and Sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day
  Least square means (LS Mean) was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline and 28 days
Population: ITT
Measure: Number; unit: Scores on a Scale
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 192 | 194 | 192
Scores on a Scale
  Baseline Least Squares Mean Symptom Score | 14.7 (0.0) | 15.5 (0.0) | 15.8 (0.0)
  Change from baseline LS Mean symptom score | -3.1 (0.0) | -3.8 (0.0) | -4.0 (0.0)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p = 0.03, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.90, 95% CI [-1.70 to -0.10]
Statistical Analysis 2: Comparison: Placebo vs Astepro 0.1%; Test type: Superiority or Other; p = 0.08, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.7, 95% CI [-1.5 to 0.1]

2. Secondary Outcome: Change From Baseline in Instantaneous Total Nasal Symprom scoreS Compared to Placebo (AM and PM Combined)and 28 Days
Description: instantaneous (subjects rate how they feel "right now") total nasal symptom score consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day.
Time Frame: baseline and 28 days
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 192 | 194 | 192
Scores on a Scale
  Baseline Symptom score | 13.28 (4.614) | 13.91 (4.616) | 14.30 (4.572)
  Overall Change from baseline | -2.72 (4.129) | -3.36 (3.898) | -3.51 (4.166)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.1%; Test type: Superiority or Other; p = 0.102, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.6419, 95% CI [-1.41 to 0.13], Standard Deviation 0.3924
Statistical Analysis 2: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p = 0.044, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.7925, 95% CI [-1.56 to -0.02], Standard Deviation 0.3935

3. Secondary Outcome: Change From Baseline in 12-hour Reflective Secondary Symptom Complex Score Compared to Placebo (AM and PM Combined)and 28 Days
Description: Reflective secondary symptom complex scores (SSCS) (post-nasal drip, itchy eyes, cough and headacdhe) were assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible SSCS score is 24 per day.
Time Frame: baseline and 28 days
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 192 | 194 | 192
Scores on a Scale
  Baseline SSCS | 11.20 (4.936) | 11.77 (5.036) | 12.39 (4.885)
  Change in baseline to Day 28 | -1.79 (3.420) | -2.23 (3.865) | -2.92 (4.053)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.1%; Change in baseline to Day 28; Test type: Superiority or Other; p = 0.226, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.4394, 95% CI [-1.15 to 0.27], Standard Deviation 0.3631
Statistical Analysis 2: Comparison: Placebo vs Astepro 0.15%; Change in baseline to Day 28; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.1252, 95% CI [-1.84 to -0.41], Standard Deviation 0.3649

4. Secondary Outcome: Change From Baseline in Rinoconjunctivitis Quality of Life Questionnaire and 28 Days
Description: A 28-item RQLQ was completed on Day 1 and Day 28 or Early temination. The RQLQ consists of 7 domains rated on a 7 point scale with 0 being not troubled by the allergy symptoms, and 6 being extremely troubled/all of the time. Domain score will be calculated from the mean score of all items in the domain. Overall score will be calculated from the mean score of all items.
Time Frame: baseline and 28 Days
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 192 | 194 | 192
Units on a Scale
  Baseline: Overall | 2.98 (1.047) | 3.18 (1.048) | 3.29 (1.091)
  Change from Baseline:Overall | -0.81 (1.112) | -1.05 (1.088) | -0.94 (1.096)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p = 0.292, ANCOVA; ANCOVA was used as a model containing treatment group and site as fixed effects with the baseline value used as covariate
Statistical Analysis 2: Comparison: Placebo vs Astepro 0.1%; Test type: Superiority or Other; p = 0.040, ANCOVA; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline on Direct Visual Nasal Exams and 28 Days
Description: Examination of head and neck (scale: None, Mild, Moderate, Severe) for Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal erythema, Mucosal Bleeding, and Crusting of mucosa. Nasal irratation was rated: 0 = None, Grade 1A = focal irritation, Grade 1B = superficial mucosal erosion, Grade 2 = moderate mucosal erosion, Grade 3 = ulceration, Grade 4 = septal perforation
Time Frame: baseline and 28 days
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 192 | 194 | 192
Participants
  Epistaxis: screening - None (n=192,197,192) | 189 | 194 | 185
  Epistaxis: screening - Mild (n=192,197,192) | 3 | 3 | 7
  Epistaxis: screening - Moderate (n=192,197,192) | 0 | 0 | 0
  Epistaxis: screening - Severe (n=192,197,192) | 0 | 0 | 0
  Epistaxis: Day 28/ET - None (n=190,192,192) | 188 | 189 | 188
  Epistaxis: Day 28/ET - Mild (n=190,192,192) | 2 | 3 | 4
  Epistaxis: Day 28/ET - Moderate (n=190,192,192) | 0 | 0 | 0
  Epistaxis: Day 28/ET - Severe (n=190,192,192) | 0 | 0 | 0
  Nasal Irritation: screening - None (n=192,197,192) | 180 | 183 | 170
  Nasal Irritationscreening Grade 1A (n=192,197,192) | 8 | 12 | 21
  Nasal Irritation screening Grade1B (n=192,197,192) | 3 | 2 | 1
  Nasal Irritationscreening Grade 2 (n=192,197,192) | 1 | 0 | 0
  Nasal Irritation screening Grade 3 (n=192,197,192) | 0 | 0 | 0
  Nasal Irritation screening Grade 4 (n=192,197,192) | 0 | 0 | 0
  Nasal Irritation Day 28/ET None (n=190,192,192) | 182 | 178 | 175
  Nasal Irritation Day 28/ETGrade 1A (n=190,192,192) | 7 | 12 | 16
  Nasal Irritation Day 28/ETGrade 1B (n=190,192,192) | 1 | 1 | 1
  Nasal Irritation Day 28/ETGrade 2 (n=190,192,192) | 0 | 0 | 0
  Nasal Irritation Day 28/ETGrade 3 (n=190,192,192) | 0 | 0 | 0
  Nasal Irritation Day 28/ETGrade 4 (n=190,192,192) | 0 | 1 | 0
  Mucosal Edema: screening - None (n=192,197,192) | 25 | 30 | 23
  Mucosal Edema: screening - Mild (n=192,197,192) | 50 | 54 | 50
  Mucosal Edema: screening Moderate (n=192,197,192) | 98 | 84 | 95
  Mucosal Edema: screening - Severe (n=192,197,192) | 19 | 29 | 24
  Mucosal Edema: Day 28/ET None (n=190,192,192) | 38 | 44 | 30
  Mucosal Edema: Day 28/ET Mild (n=190,192,192) | 69 | 71 | 71
  Mucosal Edema: Day 28/ET Moderate (n=190,192,192) | 70 | 60 | 72
  Mucosal Edema: Day 28/ET Severe (n=190,192,192) | 13 | 17 | 19
  Nasal Discharge: screening - None (n=192,197,192) | 55 | 51 | 49
  Nasal Discharge: screening - Mild (n=192,197,192) | 79 | 82 | 83
  Nasal Discharge:screening Moderate (n=192,197,192) | 48 | 51 | 49
  Nasal Discharge: screening Severe (n=192,197,192) | 10 | 13 | 11
  Nasal Discharge:Day 28/ET None (n=190,192,192) | 77 | 76 | 81
  Nasal Discharge:Day 28/ET Mild (n=190,192,192) | 75 | 85 | 72
  Nasal Discharge:Day 28/ET Moderate (n=190,192,192) | 31 | 24 | 35
  Nasal Discharge:Day 28/ET Severe (n=190,192,192) | 7 | 7 | 4
  Mucosal Erythema screening None (n=192,197,192) | 91 | 108 | 106
  Mucosal Erythema screening Mild (n=192,197,192) | 61 | 58 | 54
  Mucosal Erythema screeningModerate (n=192,197,192) | 37 | 28 | 30
  Mucosal Erythema screening Severe (n=192,197,192) | 3 | 3 | 2
  Mucosal Erythema Day 28/ET None (n=190,192,192) | 101 | 124 | 111
  Mucosal Erythema Day 28/ET Mild (n=190,192,192) | 64 | 46 | 51
  Mucosal Erythema Day 28/ET Moderate (n=190,192,192 | 23 | 20 | 26
  Mucosal Erythema Day 28/ET Severe (n=190,192,192) | 2 | 2 | 4
  Mucosal Bleeding: screening None (n=192,197,192) | 185 | 192 | 183
  Mucosal Bleeding: screening Mild (n=192,197,192) | 7 | 5 | 9
  Mucosal Bleedingscreening Moderate (n=192,197,192) | 0 | 0 | 0
  Mucosal Bleeding screening Severe (n=192,197,192) | 0 | 0 | 0
  Mucosal Bleeding: Day 28/ET None (n=190,192,192) | 189 | 189 | 184
  Mucosal Bleeding: Day 28/ET Mild (n=190,192,192) | 1 | 3 | 7
  Mucosal Bleeding Day 28/ETModerate (n=190,192,192) | 0 | 0 | 1
  Mucosal Bleeding: Day 28/ET Severe (n=190,192,192) | 0 | 0 | 0
  Crusting of Mucosa: screening None (n=192,197,192) | 173 | 178 | 173
  Crusting of Mucosa: screening Mild (n=192,197,192) | 15 | 13 | 13
  CrustingofMucosa screening Moderate(n=192,197,192) | 4 | 6 | 6
  Crusting of Mucosa screening Severe(n=192,197,192) | 0 | 0 | 0
  Crusting of Mucosa:Day 28/ET None (n=190,192,192) | 176 | 178 | 175
  Crusting of Mucosa:Day 28/ET Mild (n=190,192,192) | 14 | 12 | 16
  CrustingofMucosaDay 28/ET Moderate (n=190,192,192) | 0 | 2 | 1
  Crusting of Mucosa:Day 28/ET Severe(n=190,192,192) | 0 | 0 | 0
  Conjuntival screening None (n=192,197,192) | 126 | 145 | 134
  Conjuntival screening Mild (n=192,197,192) | 56 | 43 | 48
  Conjuntival screening Moderate n=(192,192, 192) | 10 | 9 | 10
  Conjuntival screeningSevere(n=192,197,192) | 0 | 0 | 0
  Conjuntival Day 28/ET None(n=190,192,192) | 125 | 145 | 144
  Conjuntival Day 28/ET Mild(n=190,192,192) | 57 | 34 | 36
  Conjuntival Day 28/ET Moderate(n=190,192) | 6 | 10 | 11
  Conjuntival Day 28/ET Severe (n=190,192, 192) | 2 | 3 | 1
  Erythmatous TM: screening None (n=192,197,192) | 180 | 183 | 185
  Erythmatous TM: screening Mild (n=192,197,192) | 9 | 8 | 5
  Erythmatous TM: screening Moderate(n=192,197,192) | 2 | 6 | 1
  Erythmatous TM:screening Severe (n=192,197,192) | 1 | 0 | 1
  Erythmatous TM: Day 28/ET None (n=190,192, 192) | 179 | 189 | 187
  Erythmatous TM: Day 28/ET Mild (n=190,192, 192) | 8 | 1 | 3
  Erythmatous TM: Day 28/ET Moderate (n=190,192,192) | 2 | 2 | 1
  Erythmatous TM: Day 28/ET Severe (n=190,192, 192) | 1 | 0 | 1
  Lymphadenopathy: screening None (n=192,197,192) | 186 | 189 | 188
  Lymphadenopathy: screening Mild (n=192,197,192) | 4 | 6 | 3
  Lymphadenopathy:screening Moderate (n=192,197,192) | 1 | 2 | 1
  Lymphadenopathy:screening Severe (n=192,197,192) | 1 | 0 | 0
  Lymphadenopathy: Day 28/ET None (n=190,192, 192) | 184 | 190 | 188
  Lymphadenopathy: Day 28/ET Mild (n=190,192, 192) | 5 | 1 | 3
  Lymphadenopathy Day 28/ET Moderate (n=190,192,192) | 1 | 1 | 0
  Lymphadenopathy: Day 28/ET Severe ( n=190,192,192) | 0 | 0 | 1

ADVERSE EVENTS:
Description: 0 participants were at risk for an SAE. No SAE's were observed
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/194 | 0/192
Other Adverse Events (participants affected / at risk) | 21/192 | 27/194 | 32/192
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=192) | Astepro 0.1% (N=194) | Astepro 0.15% (N=192)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 13 (13)
Dysgesusia (Nervous system disorders) | 1 (1) | 11 (11) | 9 (9)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Standard deviations for primary endpoint are not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, joint publication is required to assure that the initial publication is based on all data from all sites and investigators participating in these studies agree not to present data gathered individually or by subgroup centers before the initial publication unless jointly agreed by all other investigators and the sponsor. authorship will be determined by mutual agreement.